CLINICAL TRIAL: NCT04911686
Title: Correction of Fixed Knee Flexion Deformity in Children Distraction by Cast Wedge and Rod Lengthening
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alm-Eldeen khalf sholkamy, doctor, Assiut University
Other Study IDs: Knee flexion deformities
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-03

CONDITIONS: Flexion Deformity of Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: rod distraction — Our study entails the application of a simple method for correction of FKFD in younger children using a simple cast distraction technique. This conservative method aims at avoiding the complications of surgery in children while achieving a reasonable amount of correction.
  Other Names: hemiephysiodesis

SUMMARY:
The aim of our study is to produce gradual correction of FKFD in younger children.

DETAILED DESCRIPTION:
Management of pediatric fixed knee flexion deformities (FKFD) has always been a challenge for orthopedic surgeons. They occur due to a variety of causes, including cerebral palsy, arthrogryposis, spina bifida, trauma, and many others. The deleterious effects of FKFD include instability of gait and balance, exhaustion of extensor mechanism, and anterior knee pain, which together produce marked limitation of the activities of daily living in affected children .

Many options have been proposed for the correction of FKFD, with each having its pros and cons. Hamstring release and posterior capsulotomy are frequently used. However, extensive soft tissue release may be needed to treat severe deformities with the risk of neurovascular compromise and genu recurvatum. Supracondylar extension osteotomy with patellar tendon advancement requires postoperative non-weight bearing for at least three weeks and is associated with risk of neurovascular damage and coronal plane deformities and it is mostly used in older children and adolescent . Gradual distraction by ring fixators may be complicated by pin tract problems, fractures, and recurrence .

Our study entails the application of a simple method for correction of FKFD in younger children using a simple cast distraction technique. This conservative method aims at avoiding the complications of surgery in children while achieving a reasonable amount of correction.

ELIGIBILITY:
Inclusion Criteria:

1. Children with FKFD.
2. Age < 4 years.
3. FKFD due to congenital, traumatic, neuromuscular, infections, metabolic disorders and skeletal dysplasias.

Exclusion Criteria:

* 1. Older children less than 4 years 2. Recent Post-burn contractures and cases with unsuitable skin conditions.

Max Age: 4 Years | Sex: All
Age Groups: Child
Study Population: Children with FKFD Age < 4 years.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Correction of fixed knee flexion deformities in children using cast and rod distraction | baseline
  Amount of correction of the flexion deformity measured in degrees

SECONDARY OUTCOMES:
Correction of fixed knee flexion deformities in children using cast and rod distraction | baseline
  Rate of correction Monitor patients and report on complication like severe knee joint pain or posterior translation of tibia within the study period, pressure ulcers caused by cast indentation.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Khaled Hassan Ahmed, professor, Study Director — Analysis and interpretation of data

REFERENCES:
- [Background] Balci HI, Kocaoglu M, Eralp L, Bilen FE. Knee flexion contracture in haemophilia: treatment with circular external fixator. Haemophilia. 2014 Nov;20(6):879-83. doi: 10.1111/hae.12478. Epub 2014 Aug 21. PMID 25143070
- [Background] Spiro AS, Stenger P, Hoffmann M, Vettorazzi E, Babin K, Lipovac S, Kolb JP, Novo de Oliveira A, Rueger JM, Stuecker R. Treatment of fixed knee flexion deformity by anterior distal femoral stapling. Knee Surg Sports Traumatol Arthrosc. 2012 Dec;20(12):2413-8. doi: 10.1007/s00167-012-1915-8. Epub 2012 Feb 4. PMID 22307752